CLINICAL TRIAL: NCT01455415
Title: A Study Of Pregabalin In The Treatment Of Subjects With Painful Diabetic Peripheral Neuropathy With Background Treatment Of Nsaid For Other Pain Conditions
Brief Title: Effect Of Pregabalin Treatment In Patients With Diabetic Nerve Pain Who Currently Use A Non-Steroid Anti-Inflammatory Drug (NSAID) For Another Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: A0081268; 2011-002743-10 (EudraCT Number)
Record Dates: First submitted 2011-10-17; First posted 2011-10-20 (Estimated); Results first posted 2015-04-23 (Estimated); Last update posted 2021-01-28 (Actual); Status verified 2015-04

CONDITIONS: Painful Diabetic Peripheral Neuropathy
MeSH Terms: interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1: Pregabalin (Experimental)
  Interventions: Drug: pregabalin
- 2: Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: pregabalin — 150 - 300 mg/day in divided dose (3 time a day) for 6 weeks
  Arms: 1: Pregabalin
Drug: placebo — matching placebo 3 time a day
  Arms: 2: Placebo

SUMMARY:
This study is to test the effectiveness of pregabalin in treating nerve pain caused by diabetes. The suitable subjects will be patients who also use an non-steroid anti-inflammatory drug for another pain which is not related to the diabetic nerve pain.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 or 2 diabetes with painful neuropathy
* Currently treated with one NSAID (including COX 2 inhibitors) for a co morbid pain condition with a regular dose
* Meet pre-defined level of pain severity at entrance

Exclusion Criteria:

* History of failed pregabalin treatment due to lack of efficacy at therapeutic dose
* Participated in a previous or ongoing pregabalin clinical trial
* Neurologic disorders unrelated to diabetic neuropathy that may confound the assessment of distal neuropathic pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Actual)
Dates: Start 2011-12; Primary Completion 2013-11 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (61):
- United States (55):
  - Dedicated Clinical Research, Goodyear, Arizona
  - Clinical Research Consortium, Phoenix, Arizona
  - Arizona Research Center, Phoenix, Arizona
  - Advanced Podiatry, Phoenix, Arizona
  - Precision Trials, Phoenix, Arizona
  - The Office of Joshua D. Holland, M.D., Phoenix, Arizona
  - Genova Clinical Research, Tucson, Arizona
  - Neuro-Pain Medical Center, Fresno, California
  - Center for United Research, Inc., Lakewood, California
  - HealthCare Partners Medical Group, Los Angeles, California
  - IDS Pharmacy, Los Angeles, California
  - University of Southern California, Los Angeles, California
  - National Research Institute, Los Angeles, California
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - Coastal Connecticut Research, LLC, New London, Connecticut
  - Neurological Group, PC, New London, Connecticut
  - Chase Medical Research, LLC, Waterbury, Connecticut
  - Meridien Research, Bradenton, Florida
  - Meridien Research, Brooksville, Florida
  - Gulfcoast Clinical Research Center, Fort Myers, Florida
  - MD Clinical, Hallandale, Florida
  - AGA Clinical Trials, Hialeah, Florida
  - Palm Beach Neurological Center,, Palm Beach Gardens, Florida
  - Meridien Research, St. Petersburg, Florida
  - Meridien Research, Tampa, Florida
  - Clinical Research of Central Florida, Winter Haven, Florida
  - Columbus Research Foundation, Columbus, Georgia
  - Suburban Clinical Research, Chicago, Illinois
  - Suburban Clinical Research, Naperville, Illinois
  - Central Kentucky Research Associates, Inc., Lexington, Kentucky
  - Arthritis and Diabetes Clinic, Inc., Monroe, Louisiana
  - Beacon Clinical Research, LLC, Brockton, Massachusetts
  - Miray Medical Center, Brockton, Massachusetts
  - Genesis Clinical Research, LLC, Fall River, Massachusetts
  - Borgess Diabetes Center, Kalamazoo, Michigan
  - Borgess Research Institute, Kalamazoo, Michigan
  - Mercy Health Research, St Louis, Missouri
  - Quality Clinical Research, Inc., Omaha, Nebraska
  - Clinical Research Consortium, Las Vegas, Nevada
  - Mirkil Medical Group, Las Vegas, Nevada
  - V.Jerome Mirkil, MD, Las Vegas, Nevada
  - The Medical Research Network, LLC, New York, New York
  - Davidson Medical Ministries, Lexington, North Carolina
  - Radiant Research (admin office), Cincinnati, Ohio
  - Radiant Research, Columbus, Ohio
  - Sooner Clinical Research, Oklahoma City, Oklahoma
  - The Office of Veronique Sebastian, MD, Oklahoma City, Oklahoma
  - Sunstone Medical Research, LLC, Medford, Oregon
  - Blair Orthopedic Associates, Inc., Altoona, Pennsylvania
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Neurology and Pain Clinic, LLC, Orangeburg, South Carolina
  - New Phase Research and Development, Knoxville, Tennessee
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - Houston Neurocare, Houston, Texas
  - Centex Research, Inc., Houston, Texas
- Czechia (3):
  - UNARS, s.r.o., Pelhřimov
  - Clintrial, s.r.o., Prague
  - Fakultni nemocnice v Motole, Prague
- Fondazione PTV Policlinico Tor Vergata di Roma, Roma, Italy
- Sweden (2):
  - Center for Lakemedelsstudier, Malmo
  - Citydiabetes, Stockholm

REFERENCES:
- [Derived] Raskin P, Huffman C, Yurkewicz L, Pauer L, Scavone JM, Yang R, Parsons B. Pregabalin in Patients With Painful Diabetic Peripheral Neuropathy Using an NSAID for Other Pain Conditions: A Double-Blind Crossover Study. Clin J Pain. 2016 Mar;32(3):203-10. doi: 10.1097/AJP.0000000000000254. PMID 25968451
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0081268&StudyName=Effect%20Of%20Pregabalin%20Treatment%20In%20Patients%20With%20Diabetic%20Nerve%20Pain%20Who%20Currently%20Use%20A%20Non-Steroid%20Anti-Inflammatory%20Drug%20%28NSAID%29%20For

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 501 participants were screened, of whom 197 were withdrawn before randomization. 304 were randomized, of whom 3 discontinued before being treated. Participants were randomized at 47 centers in 3 countries: US (43), Czech Republic (3), and Italy (1). 4 centers received study drug but did not randomize participants.
Pre-assignment Details: Participants completed daily pain and sleep diary from Visit 1 (Screening) to Visit 9. Participants with a mean pain score ≥ 4 (moderate to severe pain) and those having completed ≥ 4 daily pain dairies over past 7 days and having a mean score of ≥ 4 at Visit 2 (Baseline) were randomized.
Groups:
- Pregabalin/Placebo: Participants were randomized to double-blind treatment with pregabalin for 6 weeks (150 - 300 mg/day) in period 1 followed by placebo in period 2. There was a 2-week single-blind washout (blinded to participant) between the treatment periods. A 1-week taper was administered at the end of the second treatment period, followed by a final follow-up visit.
- Placebo/Pregablin: Participants were randomized to double-blind treatment with placebo for 6 weeks in period 1 followed by pregabalin in period 2 (150 - 300 mg/day). There was a 2-week single-blind washout (blinded to participant) between the treatment periods. A 1-week taper was administered at the end of the second treatment period, followed by a final follow-up visit.
Period: Period 1
Arm/Group | Pregabalin/Placebo | Placebo/Pregablin
Started | 154 (Started=Treated) | 147 (Started=Treated)
Completed | 135 | 123
Not Completed | 19 | 24
Not completed — Adverse Event (AE) Related to Study Drug | 9 | 6
Not completed — Lost To Follow-up Related to Study Drug | 3 | 3
Not completed — Drug Error not Associated to AE | 0 | 1
Not completed — AE Not Related to Study Drug | 2 | 6
Not completed — Withdrawal by Subject | 4 | 5
Not completed — Unspecified Reason | 1 | 1
Not completed — Protocol Violation | 0 | 2
Period: Washout
Arm/Group | Pregabalin/Placebo | Placebo/Pregablin
Started | 135 | 123
Completed | 127 | 116
Not Completed | 8 | 7
Not completed — AE Related to Study Drug | 2 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Drug Error not Associated to AE | 2 | 1
Not completed — AE Not Related to Study Drug | 2 | 3
Not completed — Unspecified Reason | 1 | 2
Not completed — Protocol Violation | 0 | 1
Period: Period 2
Arm/Group | Pregabalin/Placebo | Placebo/Pregablin
Started | 127 | 116
Completed | 114 | 106
Not Completed | 13 | 10
Not completed — AE Related to Study Drug | 1 | 2
Not completed — Lost to Follow-up | 2 | 1
Not completed — AE Not Related to Study Drug | 2 | 1
Not completed — Lack of Efficacy | 2 | 0
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Unspecified Reason | 2 | 3
Not completed — Protocol Violation | 2 | 0
Period: Follow-up
Arm/Group | Pregabalin/Placebo | Placebo/Pregablin
Started | 114 | 106
Completed | 111 | 104
Not Completed | 3 | 2
Not completed — AE Related to Study Drug | 0 | 1
Not completed — Lack of Efficacy | 0 | 1
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Unspecified Reason | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat Population (ITT) included all randomized participants with at least one dose of study drug. The ITT population was analyzed according to what the randomization schedule intended for the participants to take in each period.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pregabalin/Placebo | Placebo/Pregablin | Total
Number analyzed (Participants) | 154 | 147 | 301
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.4 (9.8) | 58.4 (9.5) | 58.9 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 72 | 137
  Male | 89 | 75 | 164

OUTCOME MEASURES:

1. Secondary Outcome: Percentage of Participants Achieving 30% Reduction in Mean DPN Pain Score From Baseline at the End of Each Treatment Period (Week 6 of Each Treatment Period)
Description: Daily pain diary consisted of an 11-point numeric scale ranging from 0 ("no pain") to 10 ("worst possible pain"). Participants described their pain during the past 24 hours by having chosen the appropriate number between 0 and 10. Self assessment was performed daily in the evening before bedtime on a telephone via IVRS (time window for completion between 6.00 pm to midnight). The endpoint mean pain score was defined as the mean of the last 7 daily diary pain ratings while taking study drug in each treatment period - period 1 and period 2, respectively. A rating of 1 - 3 was considered as mild pain; 4 - 6 as moderate pain; and 7 - 10 as severe pain.
Time Frame: End of Period (includes both Visits 5 and 9)
Population: The ITT population included all randomized participants with at least one dose of study drug. The ITT population was analyzed according to what the randomization schedule intended for the participants to take in each period.
Measure: Number; unit: percentage of participants
Groups:
- Pregabalin: The below tables included data from participants while receiving pregabalin in either period of the 2-period crossover study design. This crossover study consisted of two double blind 6- week treatment periods where participants were randomized to pregabalin or placebo for the first period, and were then switched to the other treatment for the second period. There was a 2-week single-blind washout (blinded to participant) between the treatment periods. A 1-week taper was administered at the end of the second treatment period, followed by a final follow-up visit.
- Placebo: The below table included data from participants while receiving placebo in either period of the 2-period crossover study design. This crossover study consisted of two double blind 6-week treatment periods where participants were randomized to pregabalin or placebo for the first period, and were then switched to the other treatment for the second period. There was a 2-week single-blind washout (blinded to participant) between the treatment periods. A 1-week taper was administered at the end of the second treatment period, followed by a final follow-up visit.
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 272 | 276
percentage of participants | 34.56 | 31.16
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Analysis was done using a logistic regression model which included baseline pain, sequence, period and treatment as covariate; Test type: Superiority or Other; p = 0.3287, Regression, Logistic — Secondary analysis was two-sided and performed at the 0.05 significance level, without multiple comparisons' adjustment; Odds Ratio (OR) = 1.20, 95% CI 2-sided [0.83 to 1.73]

2. Secondary Outcome: Percentage of Participants Achieving 50% Reduction in Mean DPN Pain Score From Baseline at the End of Each Treatment Period (Week 6 of Each Treatment Period)
Description: as for outcome 1
Time Frame: End of Period (includes both Visits 5 and 9)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 272 | 276
percentage of participants | 20.22 | 15.58
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0625, Regression, Logistic — Secondary analysis was two-sided and performed at the 0.05 significance level, without multiple comparisons' adjustment; Odds Ratio (OR) = 1.57, 95% CI 2-sided [0.98 to 2.51]

3. Secondary Outcome: Brief Pain Inventory-Short Form (BPI-sf) Score for Pain-Severity Domain at the End of Each Treatment Period (Week 6 of Each Treatment Period)
Description: The BPI-sf is a self-administered questionnaire developed to assess the severity of pain and the impact of pain on daily functions during a 24 hour period prior to evaluation. Four items measure pain (0: no pain; 10: worst pain possible) at its "worst, "least", "average", and "now" (current pain) on an 11-point scale. Scores range from 0 - 10 with higher scores indicating greater pain severity.
Time Frame: End of Period (includes both Visits 5 and 9)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 272 | 276
units on a scale | 4.49 (0.11) | 4.48 (0.11)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Analysis was done using a linear mixed effects model which included baseline pain severity, sequence, period, and treatment as fixed effect factors and participant within sequence and within-participant error as random factors. The treatment difference (pregabalin - placebo) has been tested using within-participant variability as error term; Test type: Superiority or Other; p = 0.9448, Mixed Models Analysis — Secondary analysis was two-sided and performed at the 0.05 significance level, without multiple comparisons' adjustment; Mean Difference (Final Values) = 0.01, 95% CI 2-sided [-0.21 to 0.22], Standard Error of Mean 0.11

4. Secondary Outcome: BPI-sf Score for Pain-Interference Domain at the End of Each Treatment Period (Week 6 of Each Treatment Period)
Description: The BPI-sf is a self-administered questionnaire developed to assess the severity of pain and the impact of pain on daily functions during a 24 hour period prior to evaluation. Seven sub-questions evaluates the level of interference of pain on daily functioning (general activity, walking, work ability, mood, enjoyment of life, relations with other people, and sleep) on an 11-point scale (0: does not interfere; 10: completely interferes). Scores range from 0 - 10 with higher scores indicating greater interference.
Time Frame: End of Period (includes both Visits 5 and 9)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 272 | 276
units on a scale | 3.50 (0.12) | 3.59 (0.11)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Analysis was done using a linear mixed effects model which included baseline interference score, sequence, period, and treatment as fixed effect factors and participant within sequence and within-participant error as random factors. The treatment difference (pregabalin - placebo) has been tested using within-participant variability as error term; Test type: Superiority or Other; p = 0.4548, Mixed Models Analysis — Secondary analysis was two-sided and performed at the 0.05 significance level, without multiple comparisons' adjustment; Mean Difference (Final Values) = -0.09, 95% CI 2-sided [-0.32 to 0.14], Standard Error of Mean 0.12

5. Secondary Outcome: Mean Sleep Interference Rating Score at the End of Each Treatment Period (Week 6 of Each Treatment Period)
Description: The daily sleep diary consists of an 11-point numeric rating scale with which the participant rates how painful DPN pain has interfered with their sleep during the past 24 hours. Zero indicates "does not interfere with sleep" and 10 indicates "completely interferes (unable to sleep due to pain)". Self assessment was performed daily in the evening before bedtime on a telephone via IVRS (time window for completion between 6.00 pm to midnight) after completion of the daily pain diary.
Time Frame: End of Period (includes both Visits 5 and 9)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 272 | 276
units on a scale | 4.11 (0.12) | 4.35 (0.12)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Analysis was done using linear mixed effects model including baseline score, sequence, period, and treatment as fixed effect factors and participant within sequence and within-participant error as random factors; Test type: Superiority or Other; p = 0.0272, Mixed Models Analysis — Secondary analysis was two-sided and performed at the 0.05 significance level, without multiple comparisons' adjustment; Mean Difference (Final Values) = -0.24, 95% CI 2-sided [-0.44 to -0.03], Standard Error of Mean 0.11

6. Secondary Outcome: Hospital Anxiety and Depression Scale - Anxiety (HADS-A) Total Score at the End of Each Treatment Period (Week 6 of Each Treatment Period)
Description: The Hospital Anxiety and Depression Scale (HADS) is a 14- item self-administered questionnaire that consists of 2 scales, one measuring anxiety (HADS-A), and the other measuring depression (HADS-D). Each subscale consists of 7 statements and the participant responds as to how each item applies to him/her over the past week on 4- point response scale. Separate scores are calculated for anxiety and depression and a score (ranging from 0 to 21) is obtained for each subscale. The higher the score, the more severe the anxiety or depression.
Time Frame: End of Period (includes both Visits 5 and 9)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 272 | 276
units on a scale | 4.90 (0.18) | 4.96 (0.18)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Analysis was done using a linear mixed effects model which included baseline HADS-A score, sequence, period, and treatment as fixed effect factors and participant within sequence and within-participant error as random factors. The treatment difference (pregabalin - placebo) has been tested using within-participant variability as error term; Test type: Superiority or Other; p = 0.7344, Mixed Models Analysis — Secondary analysis was two-sided and performed at the 0.05 significance level, without multiple comparisons' adjustment; Mean Difference (Final Values) = -0.06, 95% CI 2-sided [-0.42 to 0.30], Standard Error of Mean 0.18

7. Secondary Outcome: HADS-D Total Score at the End of Each Treatment Period (Week 6 of Each Treatment Period)
Description: HADS is a 14- item self-administered questionnaire that consists of 2 scales, one measuring anxiety (HADS-A), and the other measuring depression (HADS-D). Each subscale consists of 7 statements and the participant responds as to how each item applies to him/her over the past week on 4- point response scale. Separate scores are calculated for anxiety and depression and a score (ranging from 0 to 21) is obtained for each subscale. The higher the score, the more severe the anxiety or depression.
Time Frame: End of Period (includes both Visits 5 and 9)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 272 | 276
units on a scale | 4.42 (0.17) | 4.50 (0.17)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Analysis was done using a linear mixed effects model which included baseline HADS-D score, sequence, period, and treatment as fixed effect factors and participant within sequence and within-participant error as random factors. The treatment difference (pregabalin - placebo) has been tested using within-participant variability as error term; Test type: Superiority or Other; p = 0.6007, Mixed Models Analysis — Secondary analysis was two-sided and performed at the 0.05 significance level, without multiple comparisons' adjustment; Mean Difference (Final Values) = -0.09, 95% CI 2-sided [-0.42 to 0.24], Standard Error of Mean 0.17

8. Secondary Outcome: Norfolk Quality of Life-Diabetic Neuropathy (Norfolk QOL-DN) Total Quality of Life (TQOL) Score at the End of Each Treatment Period (Week 6 of Each Treatment Period)
Description: Norfolk QOL-DN is a 35-item participant-rated questionnaire used to assess impact of diabetic neuropathy on quality of life of participants with diabetic neuropathy. All symptoms (1 - 7) are scored as either 1 or 0, indicating presence or absence of the symptom. With exception of questions 31 and 32, the other items are scored according to the 5-point Likert Scale (0 - 4, "no problem" to "severe problem"). In question 31, "good", the middle item, is scored as 0, "very good" as -1, "excellent" as -2, "fair" as 1, and "poor" as 2. In question 32, "about the same", the middle item, is scored as 0, "somewhat better" as -1, "much better" as -2, "somewhat worse" as 1, and "much worse" as 2. TQOL score should be summed as follow: sum (Σ) (1 - 7, 8 - 35). The (sub)scales are calculated without weighting of any kind, and reported as the integer sum of listed questionnaire items (range: -4 - 136). The QOL-DN version that was administered in this study was modified with a 2-week recall period.
Time Frame: End of Period (includes both Visits 5 and 9)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 272 | 276
units on a scale | 37.22 (1.03) | 38.30 (1.02)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Analysis was done using a linear mixed effects model which included baseline total score, sequence, period, and treatment as fixed effect factors and participant within sequence and within-participant error as random factors. The treatment difference (pregabalin - placebo) has been tested using within-participant variability as error term; Test type: Superiority or Other; p = 0.2987, Mixed Models Analysis — Secondary analysis was two-sided and performed at the 0.05 significance level, without multiple comparisons' adjustment; Mean Difference (Final Values) = -1.08, 95% CI 2-sided [-3.13 to 0.96], Standard Error of Mean 1.04

9. Secondary Outcome: Norfolk QOL-DN Symptoms Domain Score at the End of Each Treatment Period (Week 6 of Each Treatment Period)
Description: Norfolk QOL-DN is a 35-item participant-rated questionnaire used to assess the impact of diabetic neuropathy on quality of life of participants with diabetic neuropathy. All symptoms (1 - 7) are scored as either 1 or 0, indicating presence or absence of the symptom. Item 9 is scored according to the 5-point Likert Scale (0 - 4, "no problem" to "severe problem"). The symptoms domain score should be summed as follow: Σ (1 - 7, 9). The scales and subscales are calculated without weighting of any kind, and reported as the integer sum of the listed questionnaire items (range: 0 - 32). The QOL-DN version that was administered in this study was modified with a 2-week recall period.
Time Frame: End of Period (includes both Visits 5 and 9)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 272 | 276
units on a scale | 7.51 (0.25) | 7.86 (0.25)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Analysis was done using a linear mixed effects model which included baseline symptoms domain score, sequence, period, and treatment as fixed effect factors and participant within sequence and within-participant error as random factors. The treatment difference (pregabalin - placebo) has been tested using within-participant variability as error term; Test type: Superiority or Other; p = 0.1769, Mixed Models Analysis — Secondary analysis was two-sided and performed at the 0.05 significance level, without multiple comparisons' adjustment; Mean Difference (Final Values) = -0.35, 95% CI 2-sided [-0.85 to 0.16], Standard Error of Mean 0.26

10. Secondary Outcome: Norfolk QOL-DN Activities of Daily Living Domain Score at the End of Each Treatment Period (Week 6 of Each Treatment Period)
Description: Norfolk QOL-DN is a 35-item participant-rated questionnaire used to assess the impact of diabetic neuropathy on quality of life of participants with diabetic neuropathy. The items are scored according to the 5-point Likert Scale (0 - 4, "no problem" to "severe problem"). Activities of the daily living domain score should be summed as follow: Σ (12, 22, 23, 25, 26). Scales and subscales are calculated without weighting of any kind, and reported as integer sum of listed questionnaire items (range: 0 - 20). The QOL-DN version that was administered in the study was modified with a 2-week recall period.
Time Frame: End of Period (includes both Visits 5 and 9)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 272 | 276
units on a scale | 2.82 (0.16) | 2.94 (0.16)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Analysis was done using a linear mixed effects model which included baseline activities of daily living domain score, sequence, period, and treatment as fixed effect factors and participant within sequence and within-participant error as random factors. The treatment difference (pregabalin - placebo) has been tested using within-participant variability as error term; Test type: Superiority or Other; p = 0.5119, Mixed Models Analysis — Secondary analysis was two-sided and performed at the 0.05 significance level, without multiple comparisons' adjustment; Mean Difference (Final Values) = -0.12, 95% CI 2-sided [-0.48 to 0.24], Standard Error of Mean 0.18

11. Secondary Outcome: Norfolk QOL-DN Physical Functioning / Large Fiber Domain Score at the End of Each Treatment Period (Week 6 of Each Treatment Period)
Description: Norfolk QOL-DN is a 35-item participant-rated questionnaire used to assess the impact of diabetic neuropathy on quality of life of participants with diabetic neuropathy. With exception of questions 31 and 32, items are scored according to the 5-point Likert Scale (0 - 4, "no problem" to "severe problem"). In question 31, "good", middle item, is scored as 0, "very good" as -1 , "excellent" as -2, "fair" as 1, and "poor" as 2. In question 32, "about the same", middle item, is scored as 0, "somewhat better" as -1, "much better" as -2, "somewhat worse" as 1, and "much worse" as 2. Physical functioning / large fiber domain score should be summed as follow: Σ (8, 11, 13 - 15, 24, 27 - 35). Scales and subscales are calculated without weighting of any kind, and reported as integer sum of listed questionnaire items (range: -4 - 56). QOL-DN version that was administered in the study was modified with a 2-week recall period.
Time Frame: End of Period (includes both Visits 5 and 9)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 272 | 276
units on a scale | 23.17 (0.61) | 23.66 (0.60)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Analysis was done using a linear mixed effects model which included baseline physical functioning / large fiber domain score, sequence, period, and treatment as fixed effect factors and participant within sequence and within-participant error as random factors. The treatment difference (pregabalin - placebo) has been tested using within-participant variability as error term; Test type: Superiority or Other; p = 0.4335, Mixed Models Analysis — Secondary analysis was two-sided and performed at the 0.05 significance level, without multiple comparisons' adjustment; Mean Difference (Final Values) = -0.49, 95% CI 2-sided [-1.72 to 0.74], Standard Error of Mean 0.62

12. Secondary Outcome: Norfolk QOL-DN Small Fiber Domain Score at the End of Each Treatment Period (Week 6 of Each Treatment Period)
Description: Norfolk QOL-DN is a 35-item participant-rated questionnaire used to assess impact of diabetic neuropathy on quality of life of participants with diabetic neuropathy. The items are scored according to the 5-point Likert Scale (0 - 4, "no problem" to "severe problem"). The small fiber domain score should be summed as follow: Σ (10, 16, 17, 18). Scales and subscales are calculated without weighting of any kind, and reported as integer sum of the listed questionnaire items (range: 0 - 16). The QOL-DN version that was administered in this study was modified with a 2-week recall period.
Time Frame: End of Period (includes both Visits 5 and 9)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 272 | 276
units on a scale | 2.57 (0.16) | 2.58 (0.16)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Analysis was done using a linear mixed effects model which included baseline small fiber domain score, sequence, period, and treatment as fixed effect factors and participant within sequence and within-participant error as random factors. The treatment difference (pregabalin - placebo) has been tested using within-participant variability as error term; Test type: Superiority or Other; p = 0.9653, Mixed Models Analysis — Secondary analysis was two-sided and performed at the 0.05 significance level, without multiple comparisons' adjustment; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.31 to 0.30], Standard Error of Mean 0.16

13. Secondary Outcome: Norfolk QOL-DN Autonomic Domain Score at the End of Each Treatment Period (Week 6 of Each Treatment Period)
Description: Norfolk QOL-DN is a 35-item participant-rated questionnaire used to assess the impact of diabetic neuropathy on quality of life of participants with diabetic neuropathy. The items are scored according to the 5-point Likert Scale (0 - 4, "no problem" to "severe problem"). The autonomic domain score should be summed as follow: Σ (19, 20, 21). The scales and subscales are calculated without weighting of any kind, and reported as the integer sum of the listed questionnaire items (range: 0 - 12). The QOL-DN version that was administered in this study was modified with a 2-week recall period.
Time Frame: End of Period (includes both Visits 5 and 9)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 272 | 276
units on a scale | 1.12 (0.10) | 1.26 (0.10)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Analysis was done using a linear mixed effects model which included baseline autonomic domain score, sequence, period, and treatment as fixed effect factors and participant within sequence and within-participant error as random factors. The treatment difference (pregabalin - placebo) has been tested using within-participant variability as error term; Test type: Superiority or Other; p = 0.2690, Mixed Models Analysis — Secondary analysis was two-sided and performed at the 0.05 significance level, without multiple comparisons' adjustment; Mean Difference (Final Values) = -0.14, 95% CI 2-sided [-0.38 to 0.11], Standard Error of Mean 0.12

14. Secondary Outcome: Euro QoL-5 Dimensions (EQ-5D) Mobility Domain Score at the End of Each Treatment Period (Week 6 of Each Treatment Period)
Description: EQ-5D is a participant-completed 5-item questionnaire designed to assess health related quality of life in terms of a single index value or utility score. There are 5 dimensions: mobility, self-care, usual activities, pain / discomfort, and anxiety / depression. Each dimension is rated on a 3-point response scale (no problems, some/moderate problems, extreme problems) and the scores are combined to form a single index utility value between 0 and 1 with higher scores indicating better health.
Time Frame: End of Period (includes both Visits 5 and 9)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 272 | 276
units on a scale | 1.65 (0.03) | 1.65 (0.03)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Analysis was done using a linear mixed effects model which included baseline mobility domain score, sequence, period, and treatment as fixed effect factors and participant within sequence and within-participant error as random factors. The treatment difference (pregabalin - placebo) has been tested using within-participant variability as error term; Test type: Superiority or Other; p = 0.9951, Mixed Models Analysis — Secondary analysis was two-sided and performed at the 0.05 significance level, without multiple comparisons' adjustment; Mean Difference (Final Values) = 0.00, 95% CI 2-sided [-0.05 to 0.05], Standard Error of Mean 0.03

15. Secondary Outcome: EQ-5D Self-Care Domain Score at the End of Each Treatment Period (Week 6 of Each Treatment Period)
Description: EQ-5D is a participant-completed 5-item questionnaire designed to assess health related quality of life in terms of a single index value or utility score. There are 5 dimensions: mobility, self-care, usual activities, pain / discomfort, and anxiety / depression. Each dimension is rated on a 3-point response scale [1 = no problems, 2 = some/moderate problems, 3 = extreme problems] and the scores are combined to form a single index utility value between 0 and 1 with higher scores indicating better health.
Time Frame: End of Period (includes both Visits 5 and 9)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 272 | 276
units on a scale | 1.18 (0.02) | 1.18 (0.02)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Analysis was done using a linear mixed effects model which included baseline self-care domain score, sequence, period, and treatment as fixed effect factors and participant within sequence and within-participant error as random factors. The treatment difference (pregabalin - placebo) has been tested using within-participant variability as error term; Test type: Superiority or Other; p = 0.9726, Mixed Models Analysis — Secondary analysis was two-sided and performed at the 0.05 significance level, without multiple comparisons' adjustment; Mean Difference (Final Values) = 0.00, 95% CI 2-sided [-0.05 to 0.05], Standard Error of Mean 0.02

16. Secondary Outcome: EQ-5D Usual Activities Domain Score at the End of Each Treatment Period (Week 6 of Each Treatment Period)
Description: as for outcome 15
Time Frame: End of Period (includes both Visits 5 and 9)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 272 | 276
units on a scale | 1.53 (0.03) | 1.51 (0.03)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Analysis was done using a linear mixed effects model which included baseline usual activities domain score, sequence, period, and treatment as fixed effect factors and participant within sequence and within-participant error as random factors. The treatment difference (pregabalin - placebo) has been tested using within-participant variability as error term; Test type: Superiority or Other; p = 0.5497, Mixed Models Analysis — Secondary analysis was two-sided and performed at the 0.05 significance level, without multiple comparisons' adjustment; Mean Difference (Final Values) = 0.02, 95% CI 2-sided [-0.04 to 0.08], Standard Error of Mean 0.03

17. Secondary Outcome: EQ-5D Pain / Discomfort Domain Score at the End of Each Treatment Period (Week 6 of Each Treatment Period)
Description: as for outcome 15
Time Frame: End of Period (includes both Visits 5 and 9)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 272 | 276
units on a scale | 2.03 (0.03) | 1.98 (0.02)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Analysis was done using a linear mixed effects model which included baseline pain / discomfort domain score, sequence, period, and treatment as fixed effect factors and participant within sequence and within-participant error as random factors. The treatment difference (pregabalin - placebo) has been tested using within-participant variability as error term; Test type: Superiority or Other; p = 0.1495, Mixed Models Analysis — Secondary analysis was two-sided and performed at the 0.05 significance level, without multiple comparisons' adjustment; Mean Difference (Final Values) = 0.05, 95% CI 2-sided [-0.02 to 0.11], Standard Error of Mean 0.03

18. Secondary Outcome: EQ-5D Anxiety / Depression Domain Score at the End of Each Treatment Period (Week 6 of Each Treatment Period)
Description: as for outcome 15
Time Frame: End of Period (includes both Visits 5 and 9)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 272 | 276
units on a scale | 1.30 (0.03) | 1.35 (0.03)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Analysis was done using a linear mixed effects model which included baseline anxiety / depression domain score, sequence, period, and treatment as fixed effect factors and participant within sequence and within-participant error as random factors. The treatment difference (pregabalin - placebo) has been tested using within-participant variability as error term; Test type: Superiority or Other; p = 0.1297, Mixed Models Analysis — Secondary analysis was two-sided and performed at the 0.05 significance level, without multiple comparisons' adjustment; Mean Difference (Final Values) = -0.05, 95% CI 2-sided [-0.11 to 0.01], Standard Error of Mean 0.03

19. Secondary Outcome: EQ-5D Dolan 1997 Index Summary Score at the End of Each Treatment Period (Week 6 of Each Treatment Period)
Description: EQ-5D is a participant-completed 5-item questionnaire designed to assess health related quality of life in terms of a single index value or utility score. There are 5 dimensions: mobility, self-care, usual activities, pain / discomfort, and anxiety / depression. Each dimension is rated on a 3-point response scale [1 = no problems, 2 = some/moderate problems, 3 = extreme problems] and the scores are combined to form a single index utility value between 0 and 1 with higher scores indicating better health. The utility score is calculated using the Dolan 1997 algorithm and the revised version which was provided to the EuroQol Group by Dolan in 2001 - but later published in medical care in 2002.
Time Frame: End of Period (includes both Visits 5 and 9)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 272 | 276
units on a scale | 0.63 (0.01) | 0.65 (0.01)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Analysis was done using a linear mixed effects model which included baseline Dolan 1997 index summary score, sequence, period, and treatment as fixed effect factors and participant within sequence and within-participant error as random factors. The treatment difference (pregabalin - placebo) has been tested using within-participant variability as error term; Test type: Superiority or Other; p = 0.4279, Mixed Models Analysis — Secondary analysis was two-sided and performed at the 0.05 significance level, without multiple comparisons' adjustment; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.04 to 0.02], Standard Error of Mean 0.01

20. Secondary Outcome: EQ-5D Dolan 2002 Index Summary Score at the End of Each Treatment Period (Week 6 of Each Treatment Period)
Description: as for outcome 19
Time Frame: End of Period (includes both Visits 5 and 9)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 272 | 276
units on a scale | 0.63 (0.01) | 0.64 (0.01)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Analysis was done using a linear mixed effects model which included baseline Dolan 2001 index summary score, sequence, period, and treatment as fixed effect factors and participant within sequence and within-participant error as random factors. The treatment difference (pregabalin - placebo) has been tested using within-participant variability as error term; Test type: Superiority or Other; p = 0.5505, Mixed Models Analysis — Secondary analysis was two-sided and performed at the 0.05 significance level, without multiple comparisons' adjustment; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.04 to 0.02], Standard Error of Mean 0.01

21. Secondary Outcome: Patient Global Impression of Change (PGIC) Score at the End of Period 1 (Week 6) - Original Scores
Description: The PGIC is a participant-rated instrument that measures the participant's assessment of change in his/her overall status on a scale ranging from 1 (very much improved) to 7 (very much worse). Due to the crossover design, PGIC was analyzed at the end of period 1 (V5).
Time Frame: End of Period 1 (V5)
Population: The ITT population included all randomized participants with at least one dose of study drug. The ITT population was analyzed according to what the randomization schedule intended for the participants to take in each period. All participants who were randomized and had a period 1 PGIC value were used for this analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 148 | 143
percentage of participants
  Very much improved | 8.1 | 4.9
  Much improved | 27.7 | 19.6
  Minimally improved | 39.2 | 39.2
  No change | 14.9 | 23.1
  Minimally worse | 6.1 | 7.0
  Much worse | 2.0 | 1.4
  Very much worse | 1.4 | 2.1
  Missing | 0.7 | 2.8
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Analysis was done using a Cochran-Mantel-Haenszel (CMH) test with modified ridit transformation, under alternative hypothesis of raw mean scores differ; Test type: Superiority or Other; p = 0.0604, Cochran-Mantel-Haenszel — Secondary analysis was two-sided and performed at the 0.05 significance level, without multiple comparisons' adjustment

22. Primary Outcome: Average Diabetic Peripheral Neuropathy (DPN) Pain Based on a Numeric Rating Scale (NRS) Over the Last 7 Days of Each Treatment Period (Week 6 of Each Treatment Period)
Description: The daily pain diary consisted of an 11-point numeric scale ranging from 0 ("no pain") to 10 ("worst possible pain"). Participants described their pain during the past 24 hours by having chosen the appropriate number between 0 and 10. Self assessment was performed daily in the evening before bedtime on a telephone via interactive voice recognition system (IVRS) (time window for completion between 6.00 pm to midnight). The endpoint mean pain score was defined as the mean of the last 7 daily diary pain ratings while taking study drug in each treatment period - period 1 and period 2, respectively. A rating of 1 - 3 was considered as mild pain; 4 - 6 as moderate pain; and 7 - 10 as severe pain.
Time Frame: End of Period (includes both Visits 5 and 9)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 272 | 276
units on a scale | 4.980 (0.127) | 5.018 (0.126)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; A longitudinal analysis was done using a repeated measure linear mixed effects model including visit, treatment, an indicator variable for Week 6, and treatment by visit and by the indicator variable interaction as fixed effect factors and participant within sequence and within-participant error (estimated by using an unstructured covariance structure) as random factors. The treatment differences were tested using within-participant variability as the error term; Test type: Superiority or Other; p = 0.7174, Repeated measure mixed effects model — Primary analysis was two-sided and performed at the 0.05 significance level; The Kenward-Roger method was used to estimate denominator degrees of freedom; Mean Difference (Final Values) = -0.038, 95% CI 2-sided [-0.248 to 0.171], Standard Error of Mean 0.106

23. Secondary Outcome: PGIC Score at the End of Period 1 (Week 6) - Categorized Scores
Description: The PGIC is a participant-rated instrument that measures the participant's assessment of change in his/her overall status on a scale ranging from 1 (very much improved) to 7 (very much worse). Original scores (7 different scores) and categorized scores (4 different scores) were provided. Categorized scores were very much improved (consisting of very much improved and much improved); any improvement (consisting of very much improved, much improved, and minimally improved); no change (consisting of no change); and any worsening (consisting of minimally worse, much worse, and very much worse). Due to the crossover design, PGIC was analyzed at the end of period 1 (V5).
Time Frame: End of Period 1 (V5)
Population: as for outcome 21
Measure: Number; unit: percentage of participants
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 148 | 143
percentage of participants
  Very much/much improved | 35.8 | 24.5
  Any improvement | 75.0 | 63.6
  No change | 14.9 | 23.1
  Any worsening | 9.5 | 10.5
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Analysis was done using a CMH test with modified ridit transformation, under alternative hypothesis of raw mean scores differ; Test type: Superiority or Other; p = 0.1511, Cochran-Mantel-Haenszel — Secondary analysis was two-sided and performed at the 0.05 significance level, without multiple comparisons' adjustment

ADVERSE EVENTS:
Time Frame: From the time the participants were randomized through and including 28 calender days after the last administration of the study drug.
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study.
Arm/Group | Pregabalin | Placebo
Serious Adverse Events (participants affected / at risk) | 5/272 | 7/276
Other Adverse Events (participants affected / at risk) | 84/272 | 45/276
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin (N=272) | Placebo (N=276)
Angina pectoris (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Multi-organ failure (General disorders) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Escherichia bacteraemia (Infections and infestations) | 1 | 0
Localised infection (Infections and infestations) | 0 | 1
Lung abscess (Infections and infestations) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Ischaemic cerebral infarction (Nervous system disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin (N=272) | Placebo (N=276)
Diarrhoea (Gastrointestinal disorders) | 9 | 11
Nausea (Gastrointestinal disorders) | 9 | 8
Fatigue (General disorders) | 14 | 4
Oedema peripheral (General disorders) | 10 | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 | 5
Dizziness (Nervous system disorders) | 28 | 4
Headache (Nervous system disorders) | 9 | 8
Somnolence (Nervous system disorders) | 14 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.